CLINICAL TRIAL: NCT05015660
Title: LEFT Bundle Pacing vs Standard Right Ventricular Pacing for Heart Failure
Brief Title: Conduction System Pacing With Left Bundle Branch Pacing as Compared to Standard Right Ventricular Pacing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jacqueline Joza, Cardiac electrophysiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-7452
Record Dates: First submitted 2021-08-10; First posted 2021-08-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pacemaker DDD; Heart Block
Keywords: left bundle branch pacing
MeSH Terms: conditions — Heart Block

STUDY DESIGN:
Intervention Model Description: Prospective open-label randomized controlled trial (1:1) with blinded outcome adjudication
Who Masked: Outcomes Assessor
Masking Description: Blinded outcome adjudication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- left bundle branch pacing (Experimental)
  Interventions: Device: Left bundle branch pacing lead (Select Secure 3830 lead)
- Right ventricular pacing (Active Comparator)
  Interventions: Device: Right ventricular active fixation lead

INTERVENTIONS:
Device: Left bundle branch pacing lead (Select Secure 3830 lead) — Implantation of a left bundle branch pacing lead via sheath, to perform selective or non-selective pacing
  Arms: left bundle branch pacing
Device: Right ventricular active fixation lead — Active fixation lead (standard)
  Arms: Right ventricular pacing

SUMMARY:
High burden right ventricular (RV) pacing has been shown to increase cardiovascular mortality, incidence of heart failure (HF), worsen left ventricular (LV) function and accelerate the development of atrial fibrillation (AF). High percentage ventricular pacing and wider paced QRS in the setting of normal baseline LV ejection fractions have consistently been shown to be independent risk factors for pacing-induced cardiomyopathy. Left bundle branch pacing (LBBP) has emerged as a potential alternative pacing mechanism that may avoid LV dyssynchrony and pacing-induced LV dysfunction by mimicking native electrical conduction.

DETAILED DESCRIPTION:
We hypothesize that in patients with high degree AV block with anticipated ventricular pacing >90%, and an EF >35% patients undergoing LBBP will demonstrate a significantly lower number of the primary composite endpoint of cardiovascular death, heart failure events, and change in LVESVi as compared to standard RV pacing. Echos will be performed at baseline, 12, 24, and 36 months. NTproBNPs are performed at baseline and follow-up. There will be a core echo lab, and blinded adjudication of ECGs and events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with an ejection fraction of >35%
3. Patients with an indication for ventricular pacing and high-degree atrioventricular block where the degree of anticipated RV pacing is >90% including:

   1. Third degree AV block
   2. Symptomatic or asymptomatic second-degree AV block
   3. First degree AV block ≥ 280ms with a narrow QRS, or ≥ 240ms with an intraventricular delay (QRS duration ≥120ms)
4. Echocardiogram within the last 3 months, with ability to have DICOM images

Exclusion Criteria:

1. Indication for an implantable cardioverter defibrillator
2. Presence of a mechanical tricuspid valve
3. Any prior attempt at implantation of an ICD, CRT, HBP, or LBBP
4. Lack of capacity to consent
5. Other serious medical condition with life expectancy of <2 years
6. Pregnancy
7. Patients in whom the conduction system abnormality is expected to be transient or recover over time
8. Patients with permanent atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to cardiovascular death | 36 months
  Clinical
Time to first heart failure event | 36 months
  Defined as: (i) Emergency department (ED) visits or hospitalization for HF (requiring signs and symptoms consistent with congestive heart failure (CHF) that is responsive to oral or parenteral medications); (ii) intensification of therapy (intravenous diuretic therapy on an outpatient basis); or (iii) indication for device upgrade to CRT due to deteriorating LV function defined as an absolute decline in LVEF ≥ 10% from baseline and an LVEF ≤ 40%
Worsening LV end systolic vloume index at 2 years | 24 months
  Defined as a 15% increase from baseline on the two-year echo

SECONDARY OUTCOMES:
Cardiovascular mortality | 24 months
  CV-related
New visit for Heart Failure | 24 months
  Heart failure visit is defined as: i) Emergency department visit or hospitalization for signs and symptoms of HF that is responsive to oral or intravenous diuretics ii) intensification of therapy defined as outpatient intravenous diuretic therapy, and iii) device upgrade to cardiac resynchronization therapy.
Total mortality | 24 months
  Total mortality
Change in left ventricular ejection fraction | 24 months
  Echo parameter, change from baseline to 24 months
Change in NTproBNP level | 24 months
  From baseline to 24 months
Atrial fibrillation progression | 24 months
  Atrial fibrillation burden as noted on pacemaker
Development of new tricuspid regurgitation | 24 months
  More than mild TR from baseline
Presence of Mitral regurgitation | 24 months
  Progression/Development from baseline
Change in Lead parameter | 24 months
  stability of impedance, sensing, thresholds
Quality of Life Improvement | Evaluated at 1, 12, and 24 months, measure as compared to baseline
  Health related quality of life score: Short Form 12
Safety of procedure and long-term safety | 24 months
  Procedural and long-term safety of left bundle pacing

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre-Research Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided